CLINICAL TRIAL: NCT00584779
Title: An Open Label Pharmacokinetic Study Of Gabapentin In Japanese Subjects With Renal Impairment Including Hemodialysis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See detailed description for termination reason
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A9451160
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-10

CONDITIONS: PK Properties Of Gabapentin In Subjects With Impaired Renal Function
Keywords: Gabapentin Pharmacokinetics, renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Gabapentin
- 2 (Experimental)
  Interventions: Drug: Gabapentin
- 3 (Experimental)
  Interventions: Drug: Gabapentin
- 4 (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — CLcr:14-5 mL/min
  Arms: 3
Drug: Gabapentin — CLcr: 29-15 mL/min
  Arms: 2
Drug: Gabapentin — Hemodialysis
  Arms: 4
Drug: Gabapentin — CLcr: 29-30 mL/min
  Arms: 1

SUMMARY:
To confirm the pharmacokinetics following administration of gabapentin to Japanese subjects with renal impairment, compare the results to Western study results and confirm the adaptive possibility of dose adjustment in US package insert to Japanese.

DETAILED DESCRIPTION:
The study was terminated on September 30, 2008 at the current study site due to reported adverse events in the study subjects (n=8). While the adverse events reported were generally consistent with the known profile of gabapentin, it was decided that the study should continue at a different study site. The pharmacokinetics of gabapentin in the subjects with renal impairment will be evaluated in a separate study with a different study number at a different site. The study will be entitled: "The Pharmacokinetic Study of Gabapentin in Japanese Epileptic Subjects with Renal Impairment".

ELIGIBILITY:
Inclusion Criteria:

* The subjects whose creatinine clearance is 5-59 mL/min, or hemodialysis patients.
* The hemodialysis patients who enter this study is required hemodialysis for at least six weeks (the frequency is three times per week)

Exclusion Criteria:

* Renal allograft recipients

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | dec 2008

SECONDARY OUTCOMES:
There were no secondary outcomes measures for this study | dec 2008

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Aira-gun, Aira-cho, Kagoshima-ken, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451160&StudyName=An%20Open%20Label%20Pharmacokinetic%20Study%20Of%20Gabapentin%20%0AIn%20Japanese%20Subjects%20With%20Renal%20Impairment%0AIncluding%20Hemodialysis%0A